CLINICAL TRIAL: NCT00275275
Title: An Open Label Conversion Study of Pramipexole to Ropinirole Controlled Release (CR) in Patients With Parkinson's Disease.
Brief Title: Pramipexole Conversion to Ropinirole Controlled Release (CR)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rajesh Pahwa, MD (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor-Investigator, Rajesh Pahwa, MD, Professor and Director, Parkinson's Disease and Movement Disorder Center, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10161
Record Dates: First submitted 2006-01-09; First posted 2006-01-11 (Estimated); Results first posted 2012-08-24 (Estimated); Last update posted 2012-08-24 (Estimated); Status verified 2012-07

CONDITIONS: Parkinson Disease
Keywords: PD; Parkinson's
MeSH Terms: conditions — Parkinson Disease | interventions — ropinirole; Pramipexole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Conversion factor of Mirapex to Requip 24-Hour of 1:3. This was a switch study in which the conversion factor was being investigated to assist in the conversion from Mirapex to Requip PR. In this group, the dose of Requip PR was 3 times the dose of Mirapex.
  Interventions: Drug: Requip PR; Drug: Mirapex
- 2 (Experimental): Conversion factor of Mirapex to Requip 24-Hour of 1:4
  Interventions: Drug: Requip PR; Drug: Mirapex
- 3 (Experimental): Conversion factor of Mirapex to Requip 24-Hour of 1:5
  Interventions: Drug: Requip PR; Drug: Mirapex

INTERVENTIONS:
Drug: Requip PR — Requip 24-Hour once a day for one month
  Other Names: Requip 24-hour prolonged release (PR).
Drug: Mirapex — All subjects started the study on Mirapex. They were all then switched to Requip PR based on a conversion factor of 1:3, 1:4 or 1:5.
  Other Names: Pramipexole

SUMMARY:
A conversion study of Mirapex (pramipexole) to Requip (ropinirole) controlled release (CR) in patients with Parkinson's disease to determine the appropriate conversion ratio and side effects related to the drug.

DETAILED DESCRIPTION:
Three different arms will be used in this study. Each of the three cohorts will be treated sequentially. Each participant will be taking Mirapex for PD and will be converted to Requip CR by 1 of 3 conversion factors (mg:mg): 1:3, 1:4 and 1:5 from Mirapex to once a day Requip CR. The first five subjects of each cohort will have their initial dose administered in the clinic and be monitored for orthostatic changes. Assessments of motor function before and after conversion will be done.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Parkinson Disease
* Currently taking pramipexole
* Never have taken Requip CR

Exclusion Criteria:

* Can not have significant adverse effects to standard Requip
* Can not have atypical PD due to drugs, metabolic disorders, encephalitis or degenerative diseases
* Can not have unstable medical conditions
* Can not be taking concurrent monoamine oxidase inhibitors except for selegiline (10mg per day or less)
* Female patients of childbearing potential must be using an effective method of contraception.
* Can not be pregnant or lactating.

This may not be a complete list; there may be additional criteria which may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2006-01; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rajesh Pahwa, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled at the University of Kansas Medical Center. Enrollment started in January 2006 and ended in February 2008.
Groups:
- Mirapex to Requip 24-Hour of 1:3: Conversion factor of Mirapex to Ropinirole 24-Hour of 1:3
- Mirapex to Requip 24-Hour of 1:4: Conversion factor of Mirapex to Ropinirole 24-Hour of 1:4
- Mirapex to Requip 24-Hour of 1:5: Conversion factor of Mirapex to Ropinirole 24-Hour of 1:5
Period: Overall Study
Arm/Group | Mirapex to Requip 24-Hour of 1:3 | Mirapex to Requip 24-Hour of 1:4 | Mirapex to Requip 24-Hour of 1:5
Started | 20 | 20 | 21 (One participant was removed after enrollment and before any data was collected for him.)
Completed | 14 | 18 | 15
Not Completed | 6 | 2 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mirapex to Requip 24-Hour of 1:3 | Mirapex to Requip 24-Hour of 1:4 | Mirapex to Requip 24-Hour of 1:5 | Total
Number analyzed (Participants) | 20 | 20 | 21 | 61
Age Continuous [Mean (Standard Deviation); unit: years] | 64.1 (10.1) | 63.9 (9.7) | 66.2 (9.7) | 64.7 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 5 | 18
  Male | 12 | 15 | 16 | 43
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 21 | 61

OUTCOME MEASURES:

1. Primary Outcome: Adverse Effects Experienced
Description: Number of adverse effect experienced by participants in the different conversion ratio groups.
Time Frame: Week 4
Measure: Number; unit: number of events
Groups:
- Preferred Requip PR: This group refers to the subjects that preferred Requip PR to Mirapex
- Preferred Mirapex: This group refers to the subjects that preferred Mirapex
Arm/Group | Preferred Requip PR | Preferred Mirapex
Number analyzed (Participants) | 33 | 27
number of events | 29 | 43

2. Secondary Outcome: Number of Dose Adjustments
Description: Outcome measures the number of times a dose needed to be adjusted to compensate for adverse effects experienced.
Time Frame: Week 4
Measure: Mean (Standard Deviation); unit: number of adjustments
Groups:
- Preferred Requip PR: This is the group of subjects that preferred Requip PR to Mirapex
- Preferred Mirapex: This is the group that preferred Mirapex to Requip PR
Arm/Group | Preferred Requip PR | Preferred Mirapex
Number analyzed (Participants) | 33 | 27
number of adjustments | 0.6 (0.7) | 1.3 (1.2)

ADVERSE EVENTS:
Description: There were a total of 61 participants enrolled to the study. One participant was removed from the study before he started study related procedures. Due to that, a total of 60 participants had adverse event data recorded.
Groups:
- Preferred Requip PR: These are the subjects that preferred Requip PR to Mirapex at the end of the study
- Preferred Mirapex: These are the subjects that preferred Mirapex to Requip PR at the end of the study
Arm/Group | Preferred Requip PR | Preferred Mirapex
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/27
Other Adverse Events (participants affected / at risk) | 9/33 | 8/27
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Preferred Requip PR (N=33) | Preferred Mirapex (N=27)
PD worsening (General disorders) | 6 (6) | 8 (8)
Dizziness (General disorders) | 5 (5) | 6 (6)
Nausea (Gastrointestinal disorders) | 5 (5) | 4 (4)
Somnolence (General disorders) | 4 (4) | 5 (5)
Anxiety (General disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Edema (General disorders) | 1 (1) | 1 (1)
Headache (General disorders) | 1 (1) | 0 (0)
Heartburn (Gastrointestinal disorders) | 1 (1) | 0 (0)
Insomnia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Weakness (General disorders) | 1 (1) | 0 (0)
Confusion (General disorders) | 0 (0) | 1 (1)
Disorientation (General disorders) | 0 (0) | 1 (1)
Dyskinesia (General disorders) | 0 (0) | 2 (2)
Fatigue (General disorders) | 0 (0) | 1 (1)
Hallucinations (General disorders) | 0 (0) | 1 (1)
Leg Cramps (General disorders) | 0 (0) | 1 (1)
Slow kick in (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes